CLINICAL TRIAL: NCT06167213
Title: Safety and Effectiveness of Balloon-Expandable Bioprosthetic SAPIEN X4 Transcatheter Heart Valve - Mitral
Brief Title: ALLIANCE Mitral: Safety and Effectiveness of SAPIEN X4 Transcatheter Heart Valve - Mitral
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-05-Mitral
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease; Mitral Stenosis
Keywords: SAPIEN X4; Valve-in-Valve; Valve-in-Ring
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TMVR in failing mitral surgical bioprosthetic valve (Experimental): Transcatheter Mitral Valve Replacement (TMVR) in subjects with a failing mitral surgical bioprosthetic valve.
  Interventions: Device: SAPIEN X4 THV
- TMVR in failing native mitral valve with an annuloplasty ring (Experimental): Transcatheter Mitral Valve Replacement (TMVR) in subjects with a failing native mitral valve with an annuloplasty ring.
  Interventions: Device: SAPIEN X4 THV

INTERVENTIONS:
Device: SAPIEN X4 THV — Implantation of the SAPIEN X4 valve

SUMMARY:
This study will establish the safety and effectiveness of the Edwards SAPIEN X4 Transcatheter Heart Valve (THV) in subjects who are at high or greater surgical risk with a failing mitral surgical bioprosthetic valve or a failing native mitral valve with an annuloplasty ring.

DETAILED DESCRIPTION:
This is a prospective, single arm, multicenter, pivotal study.

ELIGIBILITY:
Inclusion Criteria:

1. Failing mitral surgical bioprosthetic valve or a failing native mitral valve with an annuloplasty ring demonstrating ≥ moderate stenosis and/or ≥ moderate insufficiency
2. Bioprosthetic surgical valve or native mitral annulus size suitable for SAPIEN X4 THV
3. NYHA functional class ≥ II
4. Heart Team agrees the subject is at high or greater surgical risk
5. The subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.

Exclusion Criteria:

1. Anatomical characteristics that would preclude safe femoral placement of the introducer sheath or safe passage of the delivery system
2. Interatrial septum or left atrium not suitable for transcatheter transseptal access
3. Failing valve has mild or greater paravalvular regurgitation
4. Failing valve is unstable, rocking, or not structurally intact
5. Annuloplasty ring dehiscence
6. Known severe patient-prosthesis mismatch or bioprosthetic valve with residual mean gradient > 10 mmHg at the end of the index procedure for implantation of the original valve
7. Annuloplasty ring type not favorable for THV implantation
8. Increased risk of THV embolization
9. Anatomical characteristics that would increase risk of left ventricular outflow tract (LVOT) obstruction
10. Surgical or transcatheter aortic valve extending into LVOT that may impinge on the mitral implant
11. Severe right ventricle (RV) dysfunction
12. Severe regurgitation or stenosis of any other valve
13. Need for aortic, tricuspid, or pulmonic valve intervention within the next 12 months
14. Left ventricular ejection fraction < 20%
15. Cardiac imaging evidence of intracardiac mass, thrombus, or vegetation
16. Myocardial infarction within 30 days prior to the study procedure
17. Hypertrophic cardiomyopathy with subvalvular obstruction
18. Subjects with planned concomitant ablation for atrial fibrillation
19. Clinically significant coronary artery disease requiring revascularization
20. Any surgical or transcatheter procedure within 30 days prior to the study procedure. Implantation of a permanent pacemaker or implantable cardioverter defibrillator (ICD) is not considered an exclusion.
21. Any planned surgical or transcatheter intervention to be performed within 30 days following the study procedure
22. Endocarditis within 180 days prior to the study procedure
23. Stroke, transient ischemic attack or neurological signs and symptoms attributed to carotid or vertebrobasilar disease within 90 days prior to the study procedure
24. Hemodynamic or respiratory instability requiring inotropic or mechanical support within 30 days prior to the study procedure
25. Renal insufficiency and/or renal replacement therapy
26. Leukopenia, anemia, thrombocytopenia
27. Inability to tolerate or condition precluding treatment with antithrombotic therapy
28. Hypercoagulable state or other condition that increases risk of thrombosis
29. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with premedication
30. Subject refuses blood products
31. Body mass index > 50 kg/m2
32. Estimated life expectancy < 24 months
33. Female who is pregnant or lactating
34. Active SARS-CoV-2 infection or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments
35. Participating in another investigational drug or device study that has not reached its primary endpoint
36. Subject considered to be part of a vulnerable population

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2038-03 (Estimated)

PRIMARY OUTCOMES:
Non-hierarchical composite of death and stroke at 1 year | 1 year
  The number of patients that died or had a stroke

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) score compared to baseline | 30 days
  The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity, and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Kansas City Cardiomyopathy Questionnaire (KCCQ) score compared to baseline | 1 year
  The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity, and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
New York Heart Association (NYHA) functional class compared to baseline | 30 days
  NYHA is a functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort.
New York Heart Association (NYHA) functional class compared to baseline | 1 year
  NYHA is a functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Krishnaswamy, MD, Principal Investigator — The Cleveland Clinic; James McCabe, MD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No